CLINICAL TRIAL: NCT05390346
Title: Screening Program of Relative Energy Deficiency in Sports in College Athletes and Establish Diagnosis and Intervention Model
Brief Title: Screening Program of Relative Energy Deficiency in Sports in College Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201902254A3
Record Dates: First submitted 2022-02-28; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-02

CONDITIONS: Relative Energy Deficiency in Sports
Keywords: Relative Energy Deficiency in Sports; Anorexia; menstrual disorder; sport injury
MeSH Terms: conditions — Anorexia; Menstruation Disturbances | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- college athletes (Experimental): Screening Program of RED-S in College Athletes and Establish Diagnosis and Intervention Model
  Interventions: Behavioral: Nutrition education

INTERVENTIONS:
Behavioral: Nutrition education — The intervention programs consist of nutrition monitoring and diet intervention.

SUMMARY:
The investigators hope that through this study will know the prevalence of Relative Energy Deficiency in Sports (RED-S) and its impact on sports injuries, performance and illness among college athletes in Taiwan. And also to find an appropriate diagnosis and intervention model to take care of athletes' health and improve sports performance Taiwan's athletes in the future.

DETAILED DESCRIPTION:
This project is divided into 3 steps for a period of two years. The first step (0-6 months) is expected to recruit a total of 100 college athletes from Taekwondo, judo, rhythmic gymnastics, and long-distance runners for Relative Energy Deficiency in Sports (RED-S) screening. The second step (7-18 months) is targeted at athletes who have been screened for potential RED-S risk (the number is tentatively 30) in the first step.

The diagnostic tools refer to the clinical assessment of Relative Energy Deficiency in Sport Clinical Assessment Tool (RED-S CAT). The third stage (19-21 months) is intervention programs targeted at the athletes who are diagnosed with RED-S (the number is tentatively 20) at 2nd step. The intervention programs consist of nutrition monitoring and diet intervention. The investigators hope that through this study will know the prevalence of RED-S and its impact on sports injuries, performance and illness among college athletes in Taiwan. And also to find an appropriate diagnosis and intervention model to take care of athletes' health and improve sports performance Taiwan's athletes in the future.

ELIGIBILITY:
Inclusion Criteria:

* (1) agree to participant this study and sign the Informed Consent Form
* (2) college athletes in National Taiwan Sport University
* (3) over the age of 18

Exclusion Criteria:

* (1) disagree to participant or unwilling to cooperate with the screening, intervention and tracking of this study
* (2) diabetes
* (3) thyroid disease
* (4) hereditary anemia
* (5) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the phenomenon of low Energy Availability (low EA) among college athletes in Taiwan. | 0-6 months
  Stage I in this study will recruit college athletes (n=100) to evaluation the subjects' energy availability (EA), calculated as energy intake (EI) minus exercise energy expenditure (EEE), normalized to fat free mass (FFM) per day (unit: kcal/kg·FFM/day). Participants' Energy Availability (EA) value lower than 30 kcal/kg·FFM/day as the status with low Energy Availability (low EA).
Stratification the risk category of RED-S of the college athletes by using the Relative Energy Deficiency in Sport Clinical Assessment Tool (RED-S CAT). | 7-18 months
  Stage II in this study will recruit the low Energy Availability (low EA) college athletes in Stage I (n=60), evaluate their risk category of RED-S by using Relative Energy Deficiency in Sport Clinical Assessment Tool (RED-S CAT).
Evaluate the improvement of energy availability (EA) after intervention with nutrition education. | 19-21 months
  Stage III in this study will recruit the low Energy Availability (low EA) college athletes in Stage II (n=40) with high or moderate risk. Evaluate the improvement of energy availability (EA) after intervention with nutrition education. Energy availability (EA), calculated as energy intake (EI) minus exercise energy expenditure (EEE), normalized to fat free mass (FFM) per day (unit: kcal/kg·FFM/day).

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Chou Lin, MD, Principal Investigator — Taoyuan Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Taoyuan Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No